CLINICAL TRIAL: NCT05775328
Title: Gender Affirmative Treatment of Hypertrichosis With Intense Pulsed Light - Effect on Hair Reduction and Quality of Life
Brief Title: Treatment of Hypertrichosis With Intense Pulsed Light
Status: Recruiting | Type: Observational
Sponsor: Alexander Shayesteh (Other Government)
Responsible Party: Sponsor-Investigator, Alexander Shayesteh, Assistant professor and senior consultant, Region Västerbotten
Organization: Region Västerbotten (Other Government)
Other Study IDs: 2023-0222-01
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Hypertrichosis; Hirsutism - Hypertrichosis
Keywords: Hypertrichosis; Hirsutism; Hair reduction; Quality of Life
MeSH Terms: conditions — Hypertrichosis; Hirsutism | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with hypertrichosis: Patients suffering from hypertrichosis or hirsutism according to Ferriman-Galway scale criteria and treated with intense pulse light for a total of 5 sessions.
  Interventions: Other: Intense pulsed light

INTERVENTIONS:
Other: Intense pulsed light — Already described in the arm/group description

SUMMARY:
The goal of this observational cohort study is to investigate the effect of intense pulsed light (IPL) for excessive hair in patients >18 years of age and in need of gender affirmative treatment, refered to the department of dermatology and venereology, Umeå University Hospital, Sweden. The main questions this study aims to answer are:

* [To evaluate the effect of consecutive IPL treatments in women with hirsutism due to polycystic ovarial syndrome (PCOS), with or without anti-androgen treatment]
* [To evaluate the effect of consecutive IPL treatments in individuals born as biologically men but in transition to become women, with or without hormonal treatment].

Patients will use self-assessed questionnaires evaluating:

* Background characteristics and time spend on concealing, reducing and treating hypertrichosis at home.
* Ferriman-Gallwey scale, regarding the intensity of their hypertrichosis.
* Dermatology Life Quality Index (DLQI) for quality of life Patients will be recruited consecutively and assessed at each visit, at the clinic before the treatments, ranging from baseline to a minimum of 5 treatment sessions.Since this is an observational study, all patients are treated by others than the researchers according to the routines och the clonic and there will be no other groups to compare the patients with.

DETAILED DESCRIPTION:
Background Hypertrichosis is defined as excessive hair in men and women while the term hirsutism is used for women with increased hair count due to hormonal changes such as increased levels of androgens. Hypertrichosis can be focal och general and hereditary or acquired. In hereditary hypertrichosis, genes or in uterus exposure to certain medications have been suggested as causes for the condition. In acquired cases, the hypertrichosis is often triggered by hormonal changes due to different medical conditions.

Investigating the cause of hypertrichosis is done by examining the patient's medical history and a complete examination of the skin. An often-used tool, for severity assessment of hypertrichosis is Ferriman & Gallwey scale. This international scale is used both by clinicians and patients for both research and in clinical practice. The Ferriman & Gallwey scale investigate 9 parts of the body with each part visually described with increasing density of hair as 4 pictures ranging from 0 point (no hair) to 4 points (dense hair). According to Ferriman & Gallwey scale, a total of ≥8 points in white and black, ≥9-10 points for mediterranean, south american and middle eastern, and ≥2 points for east Asian women indicate hypertrichosis.

Hirsutism is a common feature in women with Polycystic Ovarian Syndrome. The increased density of hair becomes noticeable during puberty and affected women report a great negative impact from the condition on their quality of life. Signs of depression and anxiety are common in women with hirsutism, due to increased social isolation and remarks regarding the hair growth and its colour by their surroundings.

Individuals with gender dysphoria and in transition of gender reassignment from the biological male sex to female, are sometimes prescribed estrogen or anti-androgens to decrease male characteristics on their body. Feminizing hormone therapy for male-to-female gender dysphoria aim to minimize body and facial hair growth. In women with mild hirsutism, there is evidence that oral contraceptives and anti-androgen treatment could be beneficial against hair growth on the body. However, the effects of these medications together with other methods such light-based treatments as intense pulsed light or lasers have not been evaluated. Intense Pulsed Light (IPL) which transmit light as energy to become absorbed as heat in the hair follicle. Repeated treatments are necessary to obtain a significant reduction of hair and long-term effects of IPL in reducing hair varies. Theoretically, the combination of anti-androgens and estrogen together with IPL, should have a synergetic effect in hair reduction no matter the intention for hair reduction. Thus, the aim of this study is to evaluate the effects of IPL, in patient with hirsutism/hypertrichosis, with or without hormonal therapy, regarding hair reduction and potential impacts on quality of life.

Materials and methods Study design Observational Cohort study Patients Patients with hirsutism and gender dysphoria are medically treated and have their follow-ups by other specialities than dermatology. However, the laser clinic at the department of dermatology and venereology, Umeå university hospital receives referrals from other departments across northern Sweden for reducing body hair in these patients. Consecutive patients referred to the department of dermatology and venereology at Umeå University Hospital due to hypertrichosis will be assessed according to our inclusion and exclusion criteria.

Inclusion criteria:18 years of age and above, diagnosis of PCOS obtained by a gynaecologist and hirsutism, diagnosis of gender dysphoria obtained after psychiatric evaluation, ≥3 points in hair density according to Ferriman-Gallwey scale on a specific part of the body. Exclusion criteria: Language barrier causing problem in understanding questionnaires or not being able to give consent, hair colours of white, orange or grey hair, skin type 5 and above according to Fitzpatrick and hereditary hypertrichosis.

Data collection The procedure of hair reduction by light based methods are done primarily by nurses and it is only in case of complications a physician is advised. Data will be collected by a coded, pre-treatment hypertrichosis specific questionnaire, asking about participants background, medical history, current medication, subjective assessment of hair density according to Visual Analogue Scale (VAS-10 point scale), localisation of hypertrichosis, Ferriman-Gallwey scale and Dermatology Life Quality Index (DLQI). DLQI is a health questionnaire for dermatology consisting of 10 questions. DLQI investigates quality of life, the duration of one week back in time. A total of 0-30 points can be yielded from the questionnaire and the more points gained, is interpreted as more negative impacts on quality of life. At each follow-up (3 months interval) the participants will be asked to fill in the questionnaire and data from a total of 5 follow-ups will be collected. All patients will be treated by nurses at the clinic, with IPL (Intense pulsed light) Nordlys by Ellipse, using a 645- to 950-nm cut off filter. Data regarding dose, wavelength and number of pulses given at each treatment session will be collected. This data is recorded and saved inside the IPL machine.

Ethical considerations All patients will be asked for their oral and written consent after receiving information about the research project. Permissions regarding questionnaires used in this study will be obtained prior to the start of the study. An ethical permission to conduct this study will be obtained from the Swedish Ethical Review Board. As this is an observational study, none of the patients will receive any other treatment than they would have for hypertrichosis, at our clinic. Participating in this study does not mean extra visits nor any conveniences for the patients other than filling out coded questionnaires at the beginning of each treatment session. The researchers in this study will not treat any of the patients. All collected data is compiled and analysed at a group level. None of data or patient characteristics will be shared with other people outside the research group and all data will be saved electronically and kept inside in a locked room.

Statistics An estimate of 32 patients is required for the study to have a 80% chance of detecting, as significant at the 5% level, a decrease in the primary outcome measure (DLQI) from 10 points to 7 points. Considering 20% lost of response/inadequate filling of questionnaires will result in a total of 39 patients needed as sample size.

Background characteristics of patients and categorical variables will be tested with Chi-test. Normally distributed and continuous data, expressed as mean and standard deviation, will be tested for significant differences with pair t-test between the treatment sessions. Non continuous data, as median and inter quartile range will be subjected to non-parametric tests such as Mann-Whitney U test. Correlations will be tested by Pearson's correlation coefficient or spearman's rank test. Bivariate logistic regression model will be used to analyse probabilities of medications such as estrogen and anti-androgens as dependent variables, tested for outcome variables such as Ferriman-Galway scale and DLQI. International Business Machines Corporation (IBM), Statistical Package for the Social Sciences (SPSS) software will be used for statistics. A p-value less ≤ 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above
* Diagnosis of PCOS obtained by a gynaecologist and hirsutism,
* Diagnosis of gender dysphoria obtained after psychiatric evaluation,
* ≥3 points in hair density according to Ferriman-Gallwey scale on a specific part of the body

Exclusion Criteria:

* Language barrier causing problem in understanding questionnaires or not being able to give consent
* Hair colours of white, orange or grey hair
* Skin type 5 and above according to Fitzpatrick
* Hereditary hypertrichosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hirsutism and gender dysphoria are medically treated and have their follow-ups by other specialities than dermatology. However, the laser clinic at the department of Dermatology and Venereology, Umeå university hospital receives referrals from other healthcare departments, across northern Sweden, for body hair reduction. Consecutive patients referred to the department of dermatology and venereology at Umeå University Hospital due to hypertrichosis will be assessed according to our inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
DLQI | 2023-2025
  The scale of Dermatology Life Quality Index. Anticipated reduction by 3 mean points between basle-line and the last treatment session.

SECONDARY OUTCOMES:
Complications | 2023-2025
  Side-effects such as pigmentation disturbances, blisters or skin shedding post-treatment. These complications will be assessed and descriptively reported.

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Nordlund, Chief, Study Director — Region Västerbotten
Locations (1):
- Norrlands University Hospital, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No
According to Swedish Law no patient data can be transferred or shared outside the location where the research is conducted. However, data on a group level can be shared upon reasonable request.

REFERENCES:
- [Background] Park AM, Khan S, Rawnsley J. Hair Biology: Growth and Pigmentation. Facial Plast Surg Clin North Am. 2018 Nov;26(4):415-424. doi: 10.1016/j.fsc.2018.06.003. Epub 2018 Aug 16. PMID 30213423
- [Background] Mimoto MS, Oyler JL, Davis AM. Evaluation and Treatment of Hirsutism in Premenopausal Women. JAMA. 2018 Apr 17;319(15):1613-1614. doi: 10.1001/jama.2018.2611. PMID 29522641
- [Background] Saleh D, Yarrarapu SNS, Cook C. Hypertrichosis. 2023 Aug 16. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK534854/ PMID 30521275
- [Background] FERRIMAN D, GALLWEY JD. Clinical assessment of body hair growth in women. J Clin Endocrinol Metab. 1961 Nov;21:1440-7. doi: 10.1210/jcem-21-11-1440. No abstract available. PMID 13892577
- [Background] DeUgarte CM, Woods KS, Bartolucci AA, Azziz R. Degree of facial and body terminal hair growth in unselected black and white women: toward a populational definition of hirsutism. J Clin Endocrinol Metab. 2006 Apr;91(4):1345-50. doi: 10.1210/jc.2004-2301. Epub 2006 Jan 31. PMID 16449347
- [Background] Escobar-Morreale HF, Carmina E, Dewailly D, Gambineri A, Kelestimur F, Moghetti P, Pugeat M, Qiao J, Wijeyaratne CN, Witchel SF, Norman RJ. Epidemiology, diagnosis and management of hirsutism: a consensus statement by the Androgen Excess and Polycystic Ovary Syndrome Society. Hum Reprod Update. 2012 Mar-Apr;18(2):146-70. doi: 10.1093/humupd/dmr042. Epub 2011 Nov 6. PMID 22064667
- [Background] Cheewadhanaraks S, Peeyananjarassri K, Choksuchat C. Clinical diagnosis of hirsutism in Thai women. J Med Assoc Thai. 2004 May;87(5):459-63. PMID 15222512
- [Background] Lindholm A, Andersson L, Eliasson M, Bixo M, Sundstrom-Poromaa I. Prevalence of symptoms associated with polycystic ovary syndrome. Int J Gynaecol Obstet. 2008 Jul;102(1):39-43. doi: 10.1016/j.ijgo.2008.01.023. Epub 2008 Mar 5. PMID 18321516
- [Background] Coffey S, Mason H. The effect of polycystic ovary syndrome on health-related quality of life. Gynecol Endocrinol. 2003 Oct;17(5):379-86. doi: 10.1080/09513590312331290268. PMID 14710585
- [Background] Clayton WJ, Lipton M, Elford J, Rustin M, Sherr L. A randomized controlled trial of laser treatment among hirsute women with polycystic ovary syndrome. Br J Dermatol. 2005 May;152(5):986-92. doi: 10.1111/j.1365-2133.2005.06426.x. PMID 15888157
- [Background] Meyer G, Boczek U, Bojunga J. Hormonal Gender Reassignment Treatment for Gender Dysphoria. Dtsch Arztebl Int. 2020 Oct 23;117(43):725-732. doi: 10.3238/arztebl.2020.0725. PMID 33559593
- [Background] van Zuuren EJ, Fedorowicz Z, Carter B, Pandis N. Interventions for hirsutism (excluding laser and photoepilation therapy alone). Cochrane Database Syst Rev. 2015 Apr 28;2015(4):CD010334. doi: 10.1002/14651858.CD010334.pub2. PMID 25918921
- [Background] Babilas P, Schreml S, Szeimies RM, Landthaler M. Intense pulsed light (IPL): a review. Lasers Surg Med. 2010 Feb;42(2):93-104. doi: 10.1002/lsm.20877. PMID 20166155
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378